CLINICAL TRIAL: NCT01379599
Title: Brief Intervention to Reduce STDs in ER Drug Users
Acronym: SAFE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Edward Bernstein, Professor of Emergency Medicine BU SOM; Professor of Community Health Sciences BUSPH, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT00218400; NCT00218400 (obsolete NCT alias)
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Sexually Transmitted Infection
Keywords: cocaine; heroin; STIs; HIV; brief motivational intervention; voluntary testing and counseling
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief motivation intervention (Experimental): Brief motivation intervention was implemented with enrollees identified with heroin and cocaine use who were allocated to the experimental group. The aim was to test the ability of a peer-delivered intervention to reduce risk of HIV and STIs related to sexual behaviors (condom use and sex while high on drugs.
  Interventions: Behavioral: brief motivation intervention
- control group (No Intervention): Care as usual.

INTERVENTIONS:
Behavioral: brief motivation intervention — Brief motivation intervention consisting of brief psychosocial counseling (20 minutes at the time of an ER visit)
  Other Names: Brief Negotiation Interview; Safe Sex: Brief Negotiation Interview (SS-BNI); motivational interviewing
  Arms: Brief motivation intervention

SUMMARY:
The goal of the proposed project is to determine the effectiveness of a brief motivational intervention among Emergency Department (ED) patients who use cocaine and/or heroin to prevent Sexually Transmitted Infections (STIs) and Human Immunodeficiency Virus (HIV) by comparing cumulative incidence and frequency of safe sex behavior between intervention and standard voluntary counseling, testing and referral to substance abuse treatment (control) groups over a one year follow-up period.

DETAILED DESCRIPTION:
Barriers to health care utilization limit drug users' interaction with the primary health care system, resulting in episodic health care received through Emergency Departments (ED) and Urgent Care Centers (UCC). Since 1994, the Boston Medical Center ED and UCC have provided substance abuse screening as standard of care. This program employs the Brief Negotiated Interview (BNI) to assess patient's reasons for drug use, readiness to change and offer intervention alternatives and referrals to substance treatment and other resources. Drug users' high rates of STIs, HIV, and Hepatitis C (HCV) and utilization of EDs and UCCs as usual sources of health care support the introduction of sexual behavior intervention in the ED and UCC setting. The proposed study will apply existing Brief Negotiation Interview (BNI) theory and research to a new behavioral context. The proposed project is a collaborative effort to adapt the BNI to encourage safe sex behaviors to prevent gonorrhea, chlamydia, and HIV among male and female ED and UCC patients age 18-54 years who use heroin and/or crack/cocaine and are not in treatment. We will enroll and 1:1 randomize 1,030 patients to intervention (safe sex BNI) or control (voluntary counseling and testing and referral to substance abuse treatment) over a 2.5-year period, with 6-month and 12-month follow-up. STIs and HIV will be diagnosed by specific laboratory assay at baseline, 6-month, and 12-month follow-up. Sexual and drug using behavior will be determined by participant self-report at baseline, 6-month, and 12-month follow-up on a 30 day time-line follow-up calender, with biochemical testing of hair samples for opiates and cocaine at enrollment and 12-month follow-up. Sexual behavior risk will be measured in terms of proportion of vaginal and anal sex acts protected by condom use and condom use at last sexual act, by sexual partner type. Differences in safe sex behavior between intervention and control groups will be evaluated using General Estimating Equation (GEE) modeling. After assessing intervention effect in the base model, we will assess intervention effect controlling for age, gender, race, injection use, HIV status and sexual and drug using behavior. An effective, brief intervention for safe sex behaviors to reduce STDs and HIV among drug users in ED and UCC settings may provide a sustainable intervention opportunity for drug users who are otherwise difficult to access.

ELIGIBILITY:
Inclusion Criteria:

* registered ER patient
* English and Spanish speakers
* 30 day use of heroin and or cocaine
* DAST score=>3

Exclusion Criteria:

* severity of medical illness
* suicidality
* police custody
* residential substance abuse treatment
* ability to provide contact information

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1030 (Actual)
Dates: Start 2004-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
unprotected sexual acts | 1 year

SECONDARY OUTCOMES:
sex acts while high on drugs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bernstein, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified may be shared on request

REFERENCES:
- [Background] Bernstein E, Heeren T, Winter M, Ashong D, Bliss C, Madico G, Ayalew B, Bernstein J. Long-term follow-up after voluntary human immunodeficiency virus/sexually transmitted infection counseling, point-of-service testing, and referral to substance abuse treatment from the emergency department. Acad Emerg Med. 2012 Apr;19(4):386-95. doi: 10.1111/j.1553-2712.2012.01314.x. PMID 22506942
- [Background] Bernstein E, Ng V, McCloskey L, Vazquez K, Ashong D, Stapleton S, Cromwell J, Bernstein J. Qualitative analysis of cocaine and heroin users' main partner sex-risk behavior: is safety in love safety in health? Addict Sci Clin Pract. 2013 Apr 23;8(1):10. doi: 10.1186/1940-0640-8-10. PMID 23618318
- [Background] Tassiopoulos K, Bernstein J, Bernstein E. Age and sharing of needle injection equipment in a cohort of Massachusetts injection drug users: an observational study. Addict Sci Clin Pract. 2013 Dec 13;8(1):20. doi: 10.1186/1940-0640-8-20. PMID 24330568
- [Background] Bernstein E, Ashong D, Heeren T, Winter M, Bliss C, Madico G, Bernstein J. The impact of a brief motivational intervention on unprotected sex and sex while high among drug-positive emergency department patients who receive STI/HIV VC/T and drug treatment referral as standard of care. AIDS Behav. 2012 Jul;16(5):1203-16. doi: 10.1007/s10461-012-0134-0. PMID 22261830